CLINICAL TRIAL: NCT06171737
Title: PCORI-CDR-2022C1-26333 Promoting Shared Decision Making for Decisions About Treatment of Severe Aortic Stenosis (IMPACT SDM Study)
Brief Title: Promoting Shared Decision Making for Severe Aortic Stenosis
Acronym: IMPACT SDM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Francisco (Other); University of Colorado, Denver (Other); University of North Carolina, Chapel Hill (Other); Emory University (Other); University of Pennsylvania (Other); University of Texas Southwestern Medical Center (Other); University of Washington (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023P001413
Record Dates: First submitted 2023-12-05; First posted 2023-12-15 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis
Keywords: aortic valve stenosis; Decision Making, Shared; decision aid; continuing medical education; cardiology; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: There is limited blinding in the trial due to the pragmatic focus and batched stepped wedge design. Patients will be told that the study is testing different types of decision support and while they will not be blinded to the materials they receive, they will not know what materials other patients receive. Clinicians and staff will be involved in delivery of the decision aids and will not be blinded to the study arm. Research staff entering survey data and conducting chart review will not be given any explicit information about study assignment; however, it is likely that they will have a sense for the arm due to the timing. The statistician conducting analyses will be blinded to group assignment at each step. For the clinician survey, we will use computer generated random assignment to select one specialist (either interventional cardiologist or cardiac surgeon) to receive the post-visit survey for each patient participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (usual care) (No Intervention): This group will receive usual care without any support for using the decision aid and without any access to the clinician training.
- Intervention (Active Comparator): The patients in this group will receive a decision aid that covers the main treatment options for aortic stenosis.
  The clinicians in this group will receive a 60-minute online training session that will provide practical tips, interactive case studies and tools for conducting shared decision making conversations covering core competencies
  Interventions: Behavioral: Decision Aid; Behavioral: Shared Decision Making Skills Training

INTERVENTIONS:
Behavioral: Decision Aid — The American College of Cardiology decision aid: Treatment Options for Severe Aortic Stenosis for patients deciding between Tavi and Surgery
  Arms: Intervention
Behavioral: Shared Decision Making Skills Training — 60-minute online training session that will provide practical tips, interactive case studies and tools for conducting shared decision making conversations covering core competencies
  Arms: Intervention

SUMMARY:
The goal of this study is to increase shared decision making for patients considering treatment for severe aortic stenosis. The main questions it aims to answer are:

* Do patient decision aids and clinician skills training course improve the quality of decisions, and do they work well for different patient populations?
* Are heart clinics able to reach the majority of patients with decision aids before their specialist visit and do the majority of clinicians complete the training course?

All participating sites will start in the usual care group and then will be randomly assigned a time to switch to the intervention group. Participants will complete surveys before and after their specialist visit.

Researchers will compare data from patients seen during usual care with data from those seen after the interventions are implemented to see if there are improvements in the quality of decisions.

DETAILED DESCRIPTION:
The goal of this study is to promote shared decision making for patients considering treatment for severe aortic stenosis. The main questions it aims to answer are:

* Do patient decision aids and clinician skills training course improve the quality of decisions, and do they work well for different patient populations?
* Are heart clinics able to reach the majority of patients with decision aids before their specialist visit and do the majority of clinicians complete the training course?

This study is a batched stepped wedge cluster randomized trial with 8 sites, about 56 surgeons and interventional cardiologists, and will enroll about 1300 patients. All participating sites will start in the usual care group and then will be randomly assigned a time to switch to the intervention group. The interventions include a patient decision aid that was created by the American College of Cardiology CardioSmart program and a online shared decision making skills training course for clinicians. The coordinating center will provide implementation support to sites when they transition to the intervention arm. Data collection is similar across usual care and intervention groups. Patient participants will complete surveys before and after their specialist visit. Clinician participants will be randomly selected to complete a survey after the patient visit. Limited clinical data will be collected from the medical record.

Researchers will compare data from patients seen during usual care with data from those seen after the interventions are implemented to see if there are improvements in the quality of decisions. Researchers will also calculate percentage of patients reached with decision aids and percentage of clinicians who complete training at each site to measure the success of the implementation.

ELIGIBILITY:
Inclusion Criteria:

* Between 65-85 years of age
* Language is English or Spanish
* Diagnosed with severe aortic stenosis defined as (e.g. an aortic valve area < 1 cm2 or as determined by clinician)
* Attend a scheduled visit with an Interventional Cardiologist and/or Cardiac Surgeon from the Heart Valve Team at a participating site

Exclusion Criteria:

* Prior aortic valve replacement surgery
* High risk for either SAVR or TAVI (e.g., Society of Thoracic Surgery score >8% or clinician determined)
* Prior coronary artery bypass surgery (CABG)
* End stage renal disease on dialysis
* Severe lung disease (chronic obstructive pulmonary disease; COPD) requiring home oxygen
* Advanced Cirrhosis
* Unable to consent for self (proxy respondents are not allowed)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Shared Decision Making | About 1 week post visit
  Shared Decision Making Process scale; Scores range 0-4 with higher scores indicating greater shared decision making occurred.

SECONDARY OUTCOMES:
Reach | About 1 week post visit
  % of eligible patients who receive decision aid
Patient Knowledge | About 1 week post visit
  Multiple choice knowledge score ranging from 0-100; higher scores indicate higher knowledge
Preference-treatment concordance | About 1 week post visit
  % of patients who received preferred treatment within 6 months of visit
Patient experience | About 1 week post visit
  CAHPS MD-patient communication subscale and visit rating score
Clinician satisfaction | About 1 week post visit
  % of clinicians who mark "very" or "extremely" satisfied with visit
Adoption | 4 weeks from the start of intervention period for each site
  % of eligible clinicians who complete the shared decision making skills training
Timeliness (time to decision) | About 1 week post visit
  % of patients who report stage of decision making is "made a decision"
Timeliness (burden) | About 1 week post visit
  % of visits where clinicians report visit length is "longer than normal"

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital; Sammy Elmariah, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - The Regents of the University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
To promote research replicability, transparency and future use of the data, de-identified data sets will be created and will be available, by request, to outside researchers. The Data Package (comprised of the de-identified Analyzable Data Set, Full Protocol, metadata, data dictionary, full statistical analysis plan, and analytic code from the project) will be deposited in the Patient-Centered Outcomes Research Institute's Data Repository at the ICPSR. Participant information sheets for the study will indicate that de-identified information will be deposited in an open access service to promote use of the data by other researchers. No information that contains identifiers or that could be used to link an individual to the data will be included in the de-identified data set. No data will be provided from qualitative transcripts as this may lead to identifying information about participants. However, codes abstracted from qualitative transcripts may be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The PCORI-designated repository will make the data available for third-party requests when PCORI makes the Final Research Report available, or at the time of publication the primary results, whichever comes first.
Access Criteria: Researchers may access the data through the PCORI-designated repository (ICPSR's website) once it is made available.

REFERENCES:
- [Derived] Sepucha K, Elmariah S, Valentine KD, Cavender MA, Chang Y, Devireddy CM, Dickert NW, Gama KD, Knoepke CE, Korngold E, Kumbhani DJ, Matlock DD, Messenger JC, Strong S, Thourani VH, Nathan A, Quader N, Brescia AA. The IMproving treatment decisions for Patients with AortiC stenosis Through Shared Decision Making (IMPACT SDM) Study: study protocol for a cluster randomized stepped wedge trial. Trials. 2024 Dec 18;25(1):820. doi: 10.1186/s13063-024-08640-6. PMID 39696639